CLINICAL TRIAL: NCT05793489
Title: Prospective Double Arm Randomized Trial for Patients With Multiple Brain Metastasis and/or Leptomeningeal Carcinomatosis: Comparison of WBRT Alone and WBRT Plus Silibinin (Sillbrain)
Brief Title: Prospective Double Arm Randomized Trial: WBRT Alone and WBRT Plus Silibinin
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Clinico Humanitas (Other)
Collaborators: health4u S.R.L (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3406
Record Dates: First submitted 2023-03-20; First posted 2023-03-31 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Brain Metastases, Adult
Keywords: Brain Metastases; WBRT; Silibinin
MeSH Terms: conditions — Brain Neoplasms | interventions — Silybin

STUDY DESIGN:
Intervention Model Description: Prospective double arm randomized trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- WBRT + Silibinin (Experimental): Patients undergo WBRT concomitant to Silibinin
  Interventions: Other: Silibinin
- WBRT (No Intervention): Patients undergo WBRT alone, total dose of 30 Gy in 10 fractions.

INTERVENTIONS:
Other: Silibinin — WBRT will be concomitant to Silibinin. Silibinin at dose of 500 mg must be administrated twice a day for the first month, after once a day continuously.
  Total dose and fractionation of WBRT: 30 Gy in 10 fractions.
  Arms: WBRT + Silibinin

SUMMARY:
The occurrence of brain metastases (BMs) is increasing given the availability of a more accurate radiological imaging such as MRI for detecting also small brain lesions and the most effective systemic therapy able to control extracranial disease. Although, the new target therapy and immunotherapy has proven to be effective on brain metastasis too, a subgroup of patients shows prove themselves unresponsive to medical treatment. A further subgroup of patients exhibit diffuse brain disease for the presence of multiple brain lesion (>10 BMs) or leptomeningeal carcinomatosis. Among these patients the most treatment employed is represented by whole brain RT. Since the 1950s, whole-brain radiation therapy (WBRT) has been the most widely used treatment for patients with multiple brain metastases, given its effectiveness in palliation, widespread availability, and ease to delivery. However, the median overall survival recorded is restricted to 3 months, on the average. A better understanding of the molecular and cellular mechanisms underlying brain metastasis might be expected to lead to improvements in the overall survival rate for these patients. Recent studies have revealed complex interactions between metastatic cancer cells and their microenvironment in the brain. Priego et al. describe that brain metastatic cells induce and maintain the co-option of a pro-metastatic program driven by signal transducer and activator of transcription 3 (STAT3) in a subpopulation of reactive astrocytes surrounding metastatic lesions. In patients, active STAT3 in reactive astrocytes correlates with reduced survival from diagnosis of intracranial metastases. Blocking STAT3 signaling in reactive astrocytes reduces experimental brain metastasis from different primary tumor sources, even at advanced stages of colonization. Silibinin (or silybin) is a natural polyphenolic flavonoid isolated from seed extracts of the herb milk thistle (Silybum marianum). Silibinin has been shown to impair STAT3 activation. Preclinical studies show that Silibinin has an anticancer effects in vitro and in vivo.

Based on this background, the investigators designed a double arm randomized trial evaluating the benefit of Silibinin (in the form of marketed supplement) associated to WBRT respect to WBRT alone.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Histological or cytological confirmation of solid tumor malignancy
* Clinical indication for whole brain radiotherapy
* Karnofsky performance status (KPS) ≥60
* Written informed consent

Exclusion Criteria:

* Prior WBRT
* KPS < 60
* Diagnosis of Lymphoproliferative disease
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2023-03-06 (Actual); Primary Completion 2025-04-04 (Actual); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 12 months
  Outcome will be evaluated in months

SECONDARY OUTCOMES:
Toxicity in term of use of corticosteroid therapy | 12 months
  Outcome will be evaluated in term of use or not of corticosteroids
Brain Distant Failure (BDF) | 12 months
  Outcome will be evaluated in months
Progression Free Survival (PFS) | 12 months
  Outcome will be evaluated in months

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Humanitas Research Hospital, Rozzano, Milano, Italy